CLINICAL TRIAL: NCT07357064
Title: Proessional Decision Making in Childbirth.
Brief Title: Professional Decision Making in Childbirth.
Acronym: PDMC
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 365059
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Childbirth Problems
Keywords: Childbirth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Midwives and obstetricians: Decision making for medical interventions in childbirth

SUMMARY:
The study is an ethnography of clinician decision making in/during childbirth for medical interventions.

DETAILED DESCRIPTION:
Medical interventions in childbirth have risen rapidly in high income countries over the last decade and this global phenomenon is reflected in the United Kingdom with, for example, caesarean section rates in England rising by 17% in the last four years to account for an average 45% of all births in 2024. Medical interventions in childbirth can be essential and have contributed to saving the lives of millions of women and children but the underpinning issues for this large rise in medical interventions in childbirth are not clear although certainly complex and multi - factorial.

The management of risk in childbirth is a central consideration as it is well documented as a key influence for professional decision making. The aim of this research study is to describe and analyse the influences on contemporary professional decisions for medical interventions in childbirth, within which risk - - how it is perceived and negotiated by clinicians and birthing parents, and the context and frameworks that support decisions to intervene or not intervene - is likely to be key.

This is a qualitative observational study with ethnography as the methodology. This approach is appropriate to explore how risk and decision making are constructed in real time contemporary frontline professional practice because it will observe what clinicians actually do (not just what they say they do) and how they create their decisions and rationales through their everyday work and professional and organisational interactions.

This research study is important because it will contribute to further understanding professional decision making for medical interventions in childbirth within a national background context of rising medical interventions, and concern about maternity care. There is not to our knowledge published qualitative research regarding this contemporary context.

This study explores professional decision making in a co - located Obstetric Unit (OU) and Alongside Midwifery Unit (AMU) in one NHS trust. A one study site is not a limitation for an in depth ethnography that will describe and analyse and the influences and complexities of contemporary clinician decision making, and from that build new insights and themes. This study as a qualitative ethnographic study will generate rich in-depth research insights that may be transferable to similar maternity settings.

ELIGIBILITY:
Inclusion Criteria:

Maternity clinicians (midwives and obstetricians, who are the clinical decision makers in childbirth)

Exclusion Criteria:

Non maternity clinicians (neonatologists, anaesthetists, maternity support workers, who may be influential to decisions made but are not the accountable decision makers)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Maternity clinicians in an NHS maternity unit
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinician decisions for medical interventions in childbirth. | From enrolment to 6 months
  This is a qualitative ethnographic study collecting qualitative data from observation and interviews with clinicians about their clinical practice and decisions for (or not for) medical interventions in childbirth. Therefore there are no specific quantitative outcome measures included. However ethnographic data will collate decisions (yes/no for medical interventions in childbirth), and code the rationales underpinning these.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Feeley, PhD, Study Director — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atkinson, P., Coffey, A., Delamont, S., Lofland, J., &Lofland, L. (2009). Handbook of Ethnography. Sage :London. Brocklehurst, P. & Kwee, A. (2011). Perinatal and maternal outcomes by planned place of birth for healthy women with low risk pregnancies: the Birthplace in England national prospective cohort study. BMJ 2011: 343: d7400 Coxon, K., Scammell, M.& Alaszewski, A. (2012). Risk, pregnancy and childbirth: What do we currently know and what do we need to know? An editorial. Health, Risk & Society. Vol 14, 2012, Issue 6, pages 503 - 510. https://doi.org/10.1080/13698575.2012.709486 Department of Health & Social Care. (2025). New Maternity Inquiry launched to Drive Improvements. Gov.uk Downe, S. & Kingdon, C. (2025).Caesareans are rising fast in the UK - but giving birth is getting worse for women. The Conversation, January 2025 Gulmezoglu, AM., Lawrie, TA., Hezelgrave, N., et al (2016). Interventions to Reduce Maternal and Newborn Morbidity and Mortality. In R. Black, R. Laxminarayan, & M. Temmerman (Eds) (2016) Maternal, Newborn and Child Health: Disease Control Priorities. 3rd Edition (Vol 2). https://www.ncbi.nih.gov/books/NBK361904/doi:10.1596?978-1-4648-0348-2_ch7 Hammersley, M. & Atkinson, P. (2019). Ethnography: Principles in Practice. Routledge: London and New York Healy, S., Humphreys, E., & Kennedy, C. (2016).Midwives' and obstetricians' perceptions of risk and its impact on clinical decision making in labour: An integrative review. Women and Birth Vol 29, Issue 2, April 2016, pages107 - 116 Healy, S., Humphreys, E., & Kennedy, C. (2017). A qualitative exploration of how midwives' and obstetricians' perception of risk affects care practices for low-risk women and normal birth. Women and Birth Vol 30, Issue 5, October 2017, pages 367-375 James, N.(1984). A postscript to nursing. In Bell, C. & Roberts, H. (Eds.) Social Researching: Politics, Problems, Practice. Routledge: London Kirkup, B. (2015). The Report of the Morecambe Bay Investigation. Indep